CLINICAL TRIAL: NCT04779684
Title: Promoting Self-determination for Institutionalized Older People Without Decision-making Capacity: Advance Care Planning by Proxy
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ralf J. Jox (Other)
Responsible Party: Sponsor-Investigator, Ralf J. Jox, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACPbp
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Advanced Dementia; Loss of Medical Decision Making Capacity
Keywords: Advance Care Planning by proxy; Surrogate decision making; Advanced Dementia; Decision making capacity

STUDY DESIGN:
Intervention Model Description: Pilot study of acceptability and fesability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACP by proxy pilot intervention group (Experimental): All participants are included in the intervention group
  Interventions: Other: Advance care planning by proxy for health care proxies of people without medical decision making capacity

INTERVENTIONS:
Other: Advance care planning by proxy for health care proxies of people without medical decision making capacity — Two discussions between a trained health professional and a health care proxy of an RACF resident who no longer has decision making capacity. First discussion focuses on life story, values, previous experiences with medical treatments, illness and death. Second discussion also includes treating physician and focuses on establishing general goals of care and medical orders in case of emergency.

SUMMARY:
This study aims to test the acceptability and feasibility of an advance care planning (ACP) intervention which has been developed to be used with the health care proxies of residential aged care facility (RACF) residents who no longer have decision making capacity for medical decisions. The intervention involves two discussions that are facilitated by a trained health professional. The first discussion aims to discuss the resident's life story, values, previous medical treatments and experiences with illness and death and whether or not they have previously documented their wishes for future care. The second discussion also involves the treating physician and aims to document anticipatory decisions for emergency situations. Follow-up discussions after 12 months or any change in situation will be conducted.

DETAILED DESCRIPTION:
Patient-centered care involves treating patients in the way that is the most aligned with their values and their self-determination. This is the aim of Advance Care Planning (ACP), a communication-based complex intervention. ACP involves accompanied reflection about one's values, anticipation of potential health problems in future states of impaired decision-making capacity, consideration of a range of treatment and care options, anticipatory decision making and the documentation and communication of these decisions to family members and health care professionals. This process ensures that a person's self-determination is respected even when she is no longer able to make health care decisions. ACP programs are well established in the English-speaking world and are currently being developed across Asia and Europe.

Participation in ACP requires decision-making capacity. Yet, many people lose this capacity before having formally expressed their care preferences. In these cases, their health care proxies, families and health professionals are called upon to make decisions on their behalf, based on what they believe the person would have wanted (presumed will). This is problematic and distressing for both family members and health professionals. The fact that many people do not participate in ACP or complete advanced directives, along with an increasing prevalence of neuro-degenerative diseases entailing a loss of decision-making capacity, means that growing numbers of people are likely to require others to make medical decisions on their behalf.

The investigator's exploratory research, confirmed by the literature, highlights an urgent unmet need for comprehensive and systematic interventions to assist in promoting self-determination of older people who lack decision making capacity. ACP by proxy (ACP-bp) has been suggested as a model to help proxies of incapacitated patients plan ahead and prepare for future care decisions. However, this model has never been specifically developed nor tested. This is why the investigators have developed a specific model of ACP-bp and aim to test it in a pilot study among proxies of residential aged care facility (RACF) residents who lack decision making capacity, primarily due to advanced dementia.

The investigators aim to test the acceptability and feasibility of this intervention and the appropriateness of outcome measures through a pilot study in two RACFs in the Swiss canton of Vaud over a period of one year. A process evaluation will be conducted through the triangulation of mixed-method data: self-report scales, semi-structured interviews, document analyses, resident health care records and an economic cost analysis. This will form the basis for a subsequent cluster-randomized control trial to test the intervention's effectiveness. This novel approach of ACP-bp has potential to promote self-determination and patient-centered care that improves both the ethical appropriateness and economic sustainability of care. It may lead to patients being treated in accordance with their wishes, reduce unnecessary overtreatment and avoid distress for family members and health care professionals. This approach also responds to calls for models of ACP which can be used in people with dementia and people living in RACFs, vulnerable populations that have generally remained invisible in ACP research so far.

ELIGIBILITY:
Health Care Proxy Inclusion Criteria:

* Is the legally authorized health care proxy for an RACF resident who: no longer has medical decision making capacity (according to medical judgement), is over 70 years of age and lives in an RACF in the canton of Vaud;
* Has sufficient language proficiency to complete a written questionnaire and participate in discussions.

Health Care Proxy Exclusion Criteria:

* Has insufficient language proficiency to complete a written questionnaire and participate in discussions.
* Lacks decision making capacity

Ages: 70 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of the ACP by proxy intervention | 12 months
  Acceptability of the intervention from the perspectives of health care proxies, RACF health professionals and physicians will be assessed through qualitative interviews asking about their experiences of the intervention. Interviews will be conducted 12 months after the start of the intervention
Feasibility of the ACP by proxy intervention in RACFs | 18 month
  Feasibility of the intervention from the perspectives of health care proxies, RACF health professionals and physicians will be assessed through qualitative interviews asking about their experiences of the intervention. Interviews will be conducted 12 months after the start of the intervention.

SECONDARY OUTCOMES:
Decisional conflict | 18 months
  Health care proxy decisional conflict in making decisions on behalf of an RACF resident who no longer has medical decision making capacity (as measured by the Decisional Conflict Scale). Higher scores indicate more decisional conflict (minimum score: 0, maximum score: 64).
Self-efficacy in giving care concordent with resident wishes | 18 months
  Health professional self-efficacy in providing care that is consistent with the wishes of a person who no longer has medical decision making capacity will be assessed through a single item numerical rating scale from 1-10 (higher scores indicate more self-efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf J Jox, MD,PhD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No